CLINICAL TRIAL: NCT03626103
Title: A Technology-Augmented Intervention to Prevent Peer Violence & Depressive Symptoms Among At-Risk Emergency Department Adolescents
Brief Title: Intervention to Prevent Peer Violence & Depressive Symptoms Among At-Risk Adolescents
Acronym: iDOVE2
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Rhode Island Hospital (Other)
Collaborators: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Prevention
Other Study IDs: R01HD093655 (NIH); R01HD093655 (NIH)
Record Dates: First submitted 2018-07-23; First posted 2018-08-10 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Depressive Disorder; Violence
Keywords: depression; violence; emergency department; mhealth; text message
MeSH Terms: conditions — Depressive Disorder; Depression; Emergencies | interventions — Communication Devices for People with Disabilities

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- + Brief ED Intervention (BI), + Text (Experimental): Participants receive both the Brief ED Intervention component (a 20-minute Motivational Interviewing- and Cognitive Behavioral Therapy-based in-Emergency Department session delivered by a bachelors'-level Research Assistant) and the Text Message Intervention component (8 weeks of an automated, tailored, two-way text-message curriculum started after the ED visit, which reinforces cognitive reappraisal, emotional regulation, and self-efficacy skills).
  Interventions: Behavioral: + Brief ED Intervention (BI); Behavioral: + Text
- + Brief ED Intervention (BI), no Text (Experimental): Participants receive the Brief ED Intervention component only (which is a 20-minute Motivational Interviewing- and Cognitive Behavioral Therapy-based in-Emergency Department session delivered by a bachelors'-level Research Assistant).
  Interventions: Behavioral: + Brief ED Intervention (BI)
- No Brief ED Intervention (BI), + Text (Experimental): Participants receive the Text Message Intervention component only (8 weeks of an automated, tailored, two-way text-message curriculum started after the ED visit, which reinforces cognitive reappraisal, emotional regulation, and self-efficacy skills). Participants receive a brochure containing online and community resources for violence and depression prevention instead of the Brief ED Intervention component.
  Interventions: Behavioral: + Text
- No Brief ED Intervention (BI), no Text (No Intervention): Participants receive neither the Brief ED Intervention component, nor the Text Message Intervention component. Participants receive a brochure containing online and community resources for violence and depression prevention, instead of the Brief ED Intervention component.

INTERVENTIONS:
Behavioral: + Brief ED Intervention (BI) — Brief ED Intervention (BI): A 20-minute Motivational Interviewing- and Cognitive Behavioral Therapy-based in-Emergency Department session delivered by a bachelors'-level Research Assistant
  Arms: + Brief ED Intervention (BI), + Text; + Brief ED Intervention (BI), no Text
Behavioral: + Text — Text: 8 weeks of an automated, tailored, two-way text-message curriculum started after the ED visit, which reinforces cognitive reappraisal, emotional regulation, and self-efficacy skills. Those that do not show improvement in mood after 7 days will be randomized into LiveText.
  Arms: + Brief ED Intervention (BI), + Text; No Brief ED Intervention (BI), + Text

SUMMARY:
The purpose of this investigation is to test the efficacy of "iDOVE2" (a brief emergency department introductory session and longitudinal automated text-message depression prevention program for high-risk teens), and to determine the most potent and parsimonious combination of intervention components for preventing peer violence and depressive symptoms among at-risk youth.

DETAILED DESCRIPTION:
Peer violence and depressive symptoms have mutual, reinforcing negative impacts on teens' emotional and behavioral regulation strategies.

The emergency department (ED) is the primary source of care for many high-risk teens. It provides an opportunity to initiate preventive interventions, to complement existing mental health treatment or to stand alone for those who may lack access to formal care. Personalized text-message interventions are accessible, feasible, and may be effective with these adolescents.

The purpose of this study is to expand on the PI's pilot randomized controlled trial (RCT) of iDOVE (K23 MH095866; PI: Ranney) by testing the efficacy of "iDOVE2" (a brief emergency department introductory session and longitudinal automated text-message depression prevention program for high-risk teens). The investigators will use a 2x2 factorial design to determine the most potent and parsimonious combination of intervention components for preventing peer violence and depressive symptoms among at-risk youth.

Participants will be identified in the course of usual clinical care in the ED. If eligible, parents will be consented and participants assented. Participants will complete a baseline assessment and will be randomized to one of four groups: Brief ED Intervention (BI) + Text; BI + No Text; No BI + Text; or No BI + No Text. Youth in the Text arm who show no signal of improvement at 7 days, per daily self-reported mood ratings, will be re-randomized to additional "LiveText" (once-weekly real-time micro-counseling via text) or to continue with standard, automated Text intervention curriculum.

At baseline and follow-ups at 2 months, 4 months, and 8 months, participants will complete assessments on depressive symptoms, violence, cognitive/behavioral skill-sets, and resource utilization.

ELIGIBILITY:
Inclusion Criteria:

* English-speaking
* presenting to the emergency department for routine care
* reporting past-year physical violence (using a modified version of The Revised Conflict Tactics Scales (CTS-2) score ≥1), as identified on a brief screen administered in the ED
* reporting past 2-week mild-to-moderate depressive symptoms (using Patient Health Questionnaire (PHQ-9) score 5-19), as identified on a brief screen administered in the ED
* Accompanied by a parent/guardian who is present and able to consent
* Possession of a cell phone with text-messaging capability

Exclusion Criteria:

* Chief complaint of suicidality, psychosis, sexual assault, or child abuse
* In police or child protective services' custody (as per state law)
* Unable to assent
* In need of emergency psychiatric care

Ages: 13 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 800 (Estimated)
Dates: Start 2018-08-01 (Actual); Primary Completion 2025-02 (Estimated); Study Completion 2025-02 (Estimated)

PRIMARY OUTCOMES:
Conflict Tactics Scale-2, physical subset (CTS-2) | Enrollment, 2 months post-enrollment, 4 months post-enrollment, 8 months post-enrollment
  Change from enrollment physical peer violence (score is summed, range 0 - 56)
Center for Epidemiologic Studies Depression Scale Revised (CESD-R) | Enrollment, 2 months post-enrollment, 4 months post-enrollment, 8 months post-enrollment
  Change from enrollment depressive symptoms (score is summed based on symptom group, range 0 - 80)

SECONDARY OUTCOMES:
Change in ED Visits for Assault-Related Injury | 12 months before enrollment and 12 months after enrollment
  Review of hospital system-wide Electronic Medical Record and state-wide Health Information Exchange to identify ED visits for peer assault
Conflict in Adolescent Dating Relationships Inventory, physical subset (CADRI) | Enrollment, 2 months post-enrollment, 4 months post-enrollment, 8 months post-enrollment
  Change from enrollment other forms of peer violence (dating relationships)
Illinois Bully Scale (IBS) | Enrollment, 2 months post-enrollment, 4 months post-enrollment, 8 months post-enrollment
  Change from enrollment other forms of peer violence (bullying)
Student School Survey | Enrollment, 2 months post-enrollment, 4 months post-enrollment, 8 months post-enrollment
  Change from enrollment other forms of peer violence (bullying)

OTHER OUTCOMES:
Self-Efficacy Questionnaire for Children (SEQ-C) | Enrollment, 2 months post-enrollment, 4 months post-enrollment, 8 months post-enrollment
  Measures emotional self-efficacy (mean score)
Emotional Regulation Questionnaire for Children and Adolescents (ERQ-CA) | Enrollment, 2 months post-enrollment, 4 months post-enrollment, 8 months post-enrollment
  Measures cognitive reappraisal (score is summed, range 6 - 30)
Bosworth Violence Self-Efficacy Scale | Enrollment, 2 months post-enrollment, 4 months post-enrollment, 8 months post-enrollment
  Measures self-rated ability to stay out of violence (mean score)

CONTACTS AND LOCATIONS:
Overall Officials: Megan L Ranney, MD MPH, Principal Investigator — Yale School of Public Health
Locations (2):
- United States (2):
  - Yale New Haven Hospital, New Haven, Connecticut
  - Rhode Island Hospital/Hasbro Children's Hospital, Providence, Rhode Island

IPD SHARING:
Plan to Share IPD: No